CLINICAL TRIAL: NCT05590611
Title: Impact of Sourdough Bread Consumption on Long-term Energy Intake: A Pilot Study of Feasibility (SOBER)
Brief Title: Impact of Sourdough Bread Consumption on Long-term Energy Intake: A Pilot Study of Feasibility
Acronym: SOBER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Full professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: S66499
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Appetite Regulation; Energy Intake; Body Weight Changes; Eating Behavior; Overweight and Obesity
MeSH Terms: conditions — Body Weight Changes; Feeding Behavior; Overweight; Obesity | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brown Bread (Placebo Comparator)
  Interventions: Other: Dietary Intervention with Brown Bread
- Wholemeal Sourdough Bread (Active Comparator)
  Interventions: Other: Dietary Intervention with Sourdough Bread

INTERVENTIONS:
Other: Dietary Intervention with Brown Bread — The participants in this group will be asked to replace all their habitual bread intake by standard brown bread. The duration of the study for each participant is 4 weeks. Apart from the change in type of bread, participants will maintain their habitual diet.
  Arms: Brown Bread
Other: Dietary Intervention with Sourdough Bread — The participants in thisgroup will be asked to replace all their habitual bread intake by wholemeal sourdough bread. The duration of the study for each participant is 4 weeks. Apart from the change in type of bread, participants will maintain their habitual diet.
  Arms: Wholemeal Sourdough Bread

SUMMARY:
The present study is a pilot study examining whether long-term sourdough bread consumption reduces energy intake and blood lipids levels over a period of 4 weeks in free-living normalweight and overweight participants.

ELIGIBILITY:
Inclusion Criteria:

* Female and male participants
* Age range 18 - 50
* BMI range >20 kg/m2 at screening visit
* Regular eating pattern (3 meals per day on at least 5 days per week)
* Habitual brown bread consumption of at least 1 slice per day (assessed by The European Prospective Investigation into Cancer (EPIC) Norfolk FFQ)
* Stable body weight for the last 6 months

Exclusion Criteria:

* Currently smoking or willingness to smoke during the study period
* Pregnancy, lactation or wish to become pregnant during the study period
* Previous or current gastrointestinal or endocrine disorders
* Previous or current substance/alcohol dependence or abuse (> 2 units per day/14 units per week)
* Coeliac disease or gluten sensitivity
* Allergy/intolerance to milk, egg, nuts, soy or sesame
* Habitual sourdough bread consumption of at least 1 slice per day (assessed by The European Prospective Investigation into Cancer (EPIC) Norfolk FFQ)
* Excessive concern about eating habits or body weight as evidenced from scores < 18 on the restraint and disinhibition subscales of the Three-Factor Eating Questionnaire (Stunkard & Messick, 1985)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Energy intake (kilocalories) | 4 weeks
  Assessed via 4-day food diaries using a mobile app

SECONDARY OUTCOMES:
Body weight | 4 weeks
Blood lipid levels | 4 weeks
  Plasma total cholesterol, triglycerides, LDL and HDL cholesterol, colourimetrically

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Verbeke, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.